CLINICAL TRIAL: NCT03303911
Title: Repeat-Dose Pharmacokinetic and Pharmacodynamic Evaluation of Cytisine in Healthy Smokers
Brief Title: A Pharmacokinetic and Pharmacodynamic Evaluation of Cytisine in Healthy Smokers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: It has been difficult to recruit participants meeting study entry criteria that are >65 years of age and not for any safety reasons.
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACH-CYT-02
Record Dates: First submitted 2017-09-28; First posted 2017-10-06 (Actual); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — cytisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cytisine 1.5 mg (Experimental): Multiple doses of 1.5 mg cytisine administered per 25-day schedule:
  * Days 1-3 (6 times daily)
  * Days 4-12 (5 times daily)
  * Days 13-16 (4 times daily)
  * Days 17-20 (3 times daily)
  * Days 21-24 (2 times daily)
  * Day 25 (Once daily)
  Interventions: Drug: Cytisine
- Cytisine 3.0 mg (Experimental): Multiple doses of 3.0 mg cytisine administered per 25-day schedule:
  * Days 1-3 (6 times daily)
  * Days 4-12 (5 times daily)
  * Days 13-16 (4 times daily)
  * Days 17-20 (3 times daily)
  * Days 21-24 (2 times daily)
  * Day 25 (Once daily)
  Interventions: Drug: Cytisine

INTERVENTIONS:
Drug: Cytisine — film-coated tablets; depending on arm assignment, 1 or 2 tablets to be taken with 240 mL water for each dose
  Other Names: Tabex

SUMMARY:
The primary objectives of this study are:

* To evaluate the pharmacokinetic (PK) parameters during repeat dosing of 1.5 mg or 3.0 mg cytisine when administered as the commercial 25-day schedule.
* To evaluate the pharmacodynamic (PD) effects (e.g., reduction in smoking) with repeat dosing of 1.5 mg or 3.0 mg cytisine when administered as the commercial 25-day schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Regular moderate cigarette smokers (minimum 10 cigarettes per day) who want to stop smoking.
2. Urine cotinine >500 ng/mL.
3. Expired air carbon monoxide (CO) > 11 parts per million (no cigarette 1 hour before test).
4. Healthy males and females 18-65+ years of age.

   1. If a female subject of child bearing potential, a negative pregnancy test at screening and admission and willing to use an effective method of contraception (unless of non-childbearing potential or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the subject) from first dose until 3 months after last dose of cytisine.
   2. If a female subject of non-child bearing potential, a negative pregnancy test at screening and admission. For the purposes of this study, this is defined as the subject being amenorrheic for at least 12 consecutive months or at least 4 months post-surgical sterilisation (including bilateral fallopian tube ligation or bilateral oophorectomy with or without hysterectomy). Menopausal status will be confirmed by demonstrating at screening that levels of follicle stimulating hormone (FSH) fall within the respective pathology reference range. In the event a subject's menopause status has been clearly established (for example, the subject indicates she has been amenorrheic for 10 years), but FSH levels are not consistent with a post-menopausal condition, determination of subject eligibility will be at Investigator's discretion following consultation with the Sponsor.
   3. If a male subject, willing to use an effective method of contraception (unless anatomically sterile or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the subject) from first dose until 3 months after last dose of cytisine.
5. Subject with no clinically significant abnormal serum biochemistry, haematology and urine examination values within 28 days before the first dose of cytisine.
6. Subject with negative urinary drugs of abuse screen, determined within 28 days before the first dose of cytisine (a positive alcohol result may be repeated at Investigator's discretion).
7. Subject with negative human immunodeficiency virus (HIV), hepatitis B surface antigen (Hep B) and hepatitis C virus antibody (Hep C) results.
8. Subject with no clinically significant abnormalities in 12-lead ECG determined after minimum of 5 minutes in supine position within 28 days before the first dose of cytisine.
9. Subject with no clinically significant abnormalities in vital signs (systolic blood pressure between 90-150 mmHg (age 18-65) and 90-160 mmHg (age >65), diastolic blood pressure (DBP) between 50 and 90 mmHg, and pulse rate (PR) between 40 110 bpm, measured on the dominant arm after minimum of 5 minutes in supine position) determined within 28 days before first dose of cytisine.
10. Subject must be available to complete the study (including in-clinic stays and post study follow-up) and comply with study restrictions.
11. Subject must provide written informed consent to participate in the study.

Exclusion Criteria:

1. Treatment with smoking cessation medications (bupropion, varenicline, any nicotine replacement therapy) within 8 weeks of first dose of cytisine.
2. Use of other forms of nicotine (e-cigarettes, smokeless tobacco) within 8 weeks of first dose of cytisine or are planning to use these products during study.
3. Known hypersensitivity/allergy reaction to varenicline, other cytisine-derivatives or any of the excipients in the Tabex formulation.
4. History of severe hypersensitivity reactions to any other drugs.
5. Current treatment with antihypertensive medicinal products, statins, tuberculostatics, cholinomimetics or anticholinesterase medicinal products.
6. History of any medical condition (e.g. gastrointestinal, renal or hepatic) or surgical condition (e.g. cholecystectomy, gastrectomy) that may affect drug pharmacokinetics (absorption, distribution, metabolism or excretion).
7. Female subjects who are breast feeding.
8. Difficulty in donating blood on either arm or known history.
9. History of alcoholism or drug abuse within last 2 years.
10. Use of non-prescription drugs, including vitamins, herbal and dietary supplements within 14 days (or 5 half-lives, whichever is longer) prior to the first dose of cytisine, unless in the opinion of the Principal Investigator the medication will not interfere with the study procedures or compromise subject safety.
11. Participated in any investigational drug clinical trial within the previous 3 months or a marketed drug trial within the previous 30 days prior to randomisation on Day 1.
12. Donation of 450 mL or more blood or had history of significant blood loss due to any reason or had plasmapheresis within 3 months before the first dose of cytisine.
13. Inability to communicate well with Principal Investigator or designees (i.e., language problem, poor mental development or impaired cerebral function).
14. Any other condition that the Principal Investigator considers making the subject unsuitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annelize Koch, MD, Principal Investigator — Simbec Research Ltd (Simbec)
Locations (1):
- Simbec Research Ltd, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (12.87) | 40.9 (12.94) | 39.0 (12.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 9 | 8 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13 | 12 | 25
  Other, Not Specified | 0 | 1 | 1
Expired Carbon Monoxide (CO) at Screening [Mean (Standard Deviation); unit: ppm] | 21.0 (8.02) | 20.7 (6.76) | 20.8 (7.27)
Urine Cotinine at Screening [Mean (Standard Deviation); unit: ng/mL] | 1661.0 (502.57) | 1944.2 (611.61) | 1802.6 (567.13)
Number of Cigarettes Smoked in the Past 24 hours on Day -1 [Mean (Standard Deviation); unit: cigarettes] | 16.31 (3.401) | 18.08 (5.171) | 17.19 (4.382)
Tobacco Craving Questionnaire - Short Form (TCQ-SF) Emotionality Score at Day -1 [Mean (Standard Deviation); unit: score on a scale] — The TCQ-SF is a 12-item questionnaire that assesses 4 components of tobacco craving: emotionality (3 items), expectancy (3 items), compulsivity (3 items) and purposefulness (3 items). Responses to each item are scored from 1 (strongly disagree) through 7 (strongly disagree). Component scores are defined as the sum of the scores within each component. The total score is defined as the sum of the 4 component scores. Emotionality scores may range from 3 to 21, with lower scores indicating weaker emotional signs of tobacco craving.
  score on a scale | 10.9 (5.25) | 11.7 (5.28) | 11.3 (5.18)
TCQ-SF Expectancy Score at Day -1 [Mean (Standard Deviation); unit: score on a scale] — The TCQ-SF is a 12-item questionnaire that assesses 4 components of tobacco craving: emotionality (3 items), expectancy (3 items), compulsivity (3 items) and purposefulness (3 items). Responses to each item are scored from 1 (strongly disagree) through 7 (strongly disagree). Component scores are defined as the sum of the scores within each component. The total score is defined as the sum of the 4 component scores. Expectancy scores may range from 3 to 21, with lower scores indicating less positive expectations about smoking.
  score on a scale | 11.4 (5.19) | 14.0 (6.47) | 12.7 (5.90)
TCQ-SF Compulsivity Score at Day -1 [Mean (Standard Deviation); unit: score on a scale] — The TCQ-SF is a 12-item questionnaire that assesses 4 components of tobacco craving: emotionality (3 items), expectancy (3 items), compulsivity (3 items) and purposefulness (3 items). Responses to each item are scored from 1 (strongly disagree) through 7 (strongly agree). Component scores are defined as the sum of the scores within each component. The total score is defined as the sum of the 4 component scores. Compulsivity scores may range from 3 to 21, with lower scores indicating compulsion to smoke was a lesser component of tobacco craving.
  score on a scale | 9.5 (4.61) | 9.5 (4.33) | 9.5 (4.38)
TCQ-SF Purposefulness Score at Day -1 [Mean (Standard Deviation); unit: score on a scale] — The TCQ-SF is a 12-item questionnaire that assesses 4 components of tobacco craving: emotionality (3 items), expectancy (3 items), compulsivity (3 items) and purposefulness (3 items). Responses to each item are scored from 1 (strongly disagree) through 7 (strongly disagree). Component scores are defined as the sum of the scores within each component. The total score is defined as the sum of the 4 component scores. Purposefulness scores may range from 3 to 21, with lower scores indicating stronger ability to not smoke.
  score on a scale | 14.9 (3.57) | 15.6 (5.27) | 15.3 (4.42)
TCQ-SF Total Score at Day -1 [Mean (Standard Deviation); unit: score on a scale] — The TCQ-SF is a 12-item questionnaire that assesses 4 components of tobacco craving: emotionality (3 items), expectancy (3 items), compulsivity (3 items) and purposefulness (3 items). Responses to each item are scored from 1 (strongly disagree) through 7 (strongly disagree). Component scores are defined as the sum of the scores within each component. The total score is defined as the sum of the 4 component scores. Total scores may range from 12 to 84, with lower scores indicating lower tobacco craving.
  score on a scale | 46.7 (12.96) | 50.8 (16.89) | 48.7 (14.90)
Fagerström Test for Nicotine Dependence Total Score at Day -1 [Mean (Standard Deviation); unit: score on a scale] — The Fagerström Nicotine Dependence Questionnaire (FTND) is a measure of nicotine dependence. The FTND total score is defined as the sum of the scores from 6 questions, provided all 6 questions have been completed. The FTND responses are assigned numerical values. Total Scores may range from 1 to10, with lower scores indicating less dependence on nicotine..
  score on a scale | 4.7 (1.60) | 5.3 (1.38) | 5.0 (1.50)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: after the first dose and the last dose on Day 1; after the last dose on Days 2, 3, 12, 16, 20, 24; and after the morning dose on Day 25
Population: Pharmacokinetic (PK) Set: All randomized participants who completed all cytisine dosing on Days 1-3, completed >90% cytisine dosing on Days 4-25 and complied with protocol-specified criteria. Participants with an assessment at given timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 13 | 13
ng/mL
  Day 1, first dose | 21.1 (24.8) | 40.0 (26.8)
  Day 1, last dose | 33.8 (20.0) | 81.4 (30.1)
  Day 2, last dose | 32.9 (22.3) | 85.1 (20.9)
  Day 3, last dose | 35.9 (21.7) | 88.1 (19.3)
  Day 12, last dose | 29.9 (24.9) | 69.9 (31.5)
  Day 16, last dose | 23.7 (31.4) | 50.5 (26.5)
  Day 20, last dose: number analyzed (Participants) | 12 | 13
  Day 20, last dose | 23.0 (22.1) | 49.7 (30.9)
  Day 24, last dose: number analyzed (Participants) | 12 | 13
  Day 24, last dose | 16.0 (28.3) | 42.0 (33.6)
  Day 25: number analyzed (Participants) | 12 | 13
  Day 25 | 12.6 (19.4) | 28.1 (27.4)

2. Primary Outcome: Time of Occurrence of Cmax (Tmax)
Time Frame: as for outcome 1
Population: PK Set: All randomized participants who completed all cytisine dosing on Days 1-3, completed >90% cytisine dosing on Days 4-25 and complied with protocol-specified criteria. Participants with an assessment at given time point.
Measure: Median (Full Range); unit: hours
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 13 | 13
hours
  Day 1, first dose | 0.500 [0.500 to 0.750] | 0.750 [0.500 to 1.00]
  Day 1, last dose | 1.00 [0.00 to 2.50] | 1.00 [0.00 to 2.50]
  Day 2, last dose | 1.00 [0.00 to 3.50] | 1.00 [0.00 to 3.50]
  Day 3, last dose | 1.00 [0.500 to 3.00] | 1.00 [0.00 to 2.03]
  Day 12, last dose | 1.00 [0.00 to 3.05] | 1.02 [0.00 to 2.00]
  Day 16, last dose | 2.50 [0.00 to 4.02] | 2.00 [1.00 to 6.50]
  Day 20, last dose: number analyzed (Participants) | 12 | 13
  Day 20, last dose | 1.50 [1.00 to 5.50] | 1.00 [0.00 to 6.50]
  Day 24, last dose: number analyzed (Participants) | 12 | 13
  Day 24, last dose | 2.00 [1.00 to 4.00] | 1.00 [1.00 to 3.00]
  Day 25: number analyzed (Participants) | 12 | 13
  Day 25 | 2.50 [0.500 to 5.00] | 2.25 [0.500 to 3.75]

3. Primary Outcome: Minimum Observed Plasma Concentration (Cmin)
Time Frame: after the first dose on Days 4, 13, 17, 21 and 25
Population: PK Set: All randomized participants who completed all cytisine dosing on Days 1-3, completed >90% cytisine dosing on Days 4-25 and complied with protocol-specified criteria. Participants with an assessment at given timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 13 | 13
ng/mL
  Day 4, first dose | 5.36 (47.7) | 13.2 (27.4)
  Day 13, first dose | 5.16 (48.2) | 12.6 (33.0)
  Day 17, first dose | 4.19 (64.7) | 8.50 (38.3)
  Day 21, first dose | 3.13 (83.4) | 6.34 (39.0)
  Day 25: number analyzed (Participants) | 12 | 13
  Day 25 | 3.16 (188.9) | 3.74 (42.4)

4. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) From Time Zero to the Last Sampling Time (AUC0-t)
Time Frame: after the administration of the final dose of cytisine on Day 25
Population: PK Set: All randomized participants who completed all cytisine dosing on Days 1-3, completed >90% cytisine dosing on Days 4-25 and complied with protocol-specified criteria. Participants with an assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 12 | 13
h*ng/mL | 67.0 (27.4) | 185 (32.3)

5. Primary Outcome: Total AUC From Time Zero to Infinity (AUC0-∞)
Time Frame: after the administration of the final dose of cytisine on Day 25
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 12 | 13
h*ng/mL | 82.6 (30.4) | 213 (28.0)

6. Primary Outcome: Residual Area or Percentage of Extrapolated Part for the Calculation of AUC0-∞ (%AUC)
Time Frame: after the administration of the final dose of cytisine on Day 25
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of extrapolated part
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 12 | 13
percentage of extrapolated part | 18.0 (28.9) | 11.7 (40.1)

7. Primary Outcome: Apparent Terminal Elimination Rate Constant (λz)
Time Frame: after the administration of the final dose of cytisine on Day 25
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 12 | 13
1/hour | 0.185 (26.4) | 0.152 (16.9)

8. Primary Outcome: Apparent Terminal Elimination Half-Life (t1/2)
Time Frame: after the administration of the final dose of cytisine on Day 25
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 12 | 13
hours | 3.75 (24.7) | 4.57 (17.2)

9. Primary Outcome: Number of Cigarettes Smoked Daily During Treatment and at Day 26
Time Frame: Day 1 through Day 26
Population: Pharmacodynamic (PD) Set: All participants in the PK set who had an available baseline result and at least 1 on-treatment result with regards to urine cotinine, expired air CO or daily cigarette consumption and did not incur a major protocol deviation. Participants with a valid assessment at given time point.
Measure: Mean (Standard Deviation); unit: cigarettes smoked in the past 24 hours
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 13 | 13
cigarettes smoked in the past 24 hours
  Day -1 | 16.31 (3.401) | 18.08 (5.171)
  Day 1 | 7.31 (6.088) | 8.77 (6.882)
  Day 2 | 3.69 (1.437) | 4.08 (1.801)
  Day 3: number analyzed (Participants) | 11 | 13
  Day 3 | 4.00 (1.673) | 4.46 (1.854)
  Day 4 | 4.77 (2.682) | 6.15 (3.555)
  Day 5 | 4.08 (2.629) | 5.69 (3.568)
  Day 6 | 4.85 (3.826) | 7.00 (4.778)
  Day 7 | 4.19 (4.018) | 4.85 (4.180)
  Day 8 | 4.15 (3.760) | 5.38 (4.073)
  Day 9 | 4.77 (4.438) | 5.08 (4.555)
  Day 10 | 4.62 (4.234) | 4.54 (4.557)
  Day 11 | 3.81 (3.497) | 4.62 (4.292)
  Day 12 | 3.31 (3.545) | 3.69 (3.637)
  Day 13 | 4.15 (4.038) | 5.00 (4.163)
  Day 14 | 4.00 (3.786) | 3.69 (4.535)
  Day 15 | 4.23 (3.876) | 3.62 (4.331)
  Day 16 | 3.85 (3.648) | 3.08 (3.451)
  Day 17 | 4.00 (4.163) | 3.77 (4.781)
  Day 18 | 3.69 (3.903) | 3.92 (4.873)
  Day 19 | 3.69 (3.881) | 3.54 (4.789)
  Day 20: number analyzed (Participants) | 12 | 13
  Day 20 | 3.25 (3.671) | 2.58 (3.528)
  Day 21 | 4.54 (4.719) | 2.92 (4.462)
  Day 22 | 4.00 (4.163) | 3.00 (3.958)
  Day 23 | 4.38 (4.407) | 2.69 (4.151)
  Day 24 | 3.08 (2.985) | 2.38 (3.042)
  Day 25: number analyzed (Participants) | 12 | 13
  Day 25 | 1.17 (1.467) | 0.85 (1.214)
  Day 26 | 4.23 (4.206) | 3.00 (4.778)

10. Primary Outcome: Change From Baseline in Number of Cigarettes Smoked Daily up to Day 26
Time Frame: Baseline, Day 1 through Day 26
Population: PD Set: All participants in the PK set who had an available baseline result and at least 1 on-treatment result with regards to urine cotinine, expired air CO or daily cigarette consumption and did not incur a major protocol deviation. Participants with a valid assessment at given time point.
Measure: Mean (Standard Deviation); unit: cigarettes smoked in the past 24 hours
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 13 | 13
cigarettes smoked in the past 24 hours
  Day 1 | -9.00 (5.745) | -9.31 (7.169)
  Day 2 | -12.62 (3.664) | -14.00 (5.000)
  Day 3: number analyzed (Participants) | 11 | 13
  Day 3 | -11.91 (3.885) | -13.62 (5.723)
  Day 4 | -11.54 (4.737) | -11.92 (6.144)
  Day 5 | -12.23 (4.475) | -12.38 (5.665)
  Day 6 | -11.46 (4.371) | -11.08 (7.005)
  Day 7 | -12.12 (4.718) | -13.23 (5.388)
  Day 8 | -12.15 (4.580) | -12.69 (5.391)
  Day 9 | -11.54 (5.333) | -13.00 (5.845)
  Day 10 | -11.69 (4.697) | -13.54 (5.425)
  Day 11 | -12.50 (4.173) | -13.46 (4.789)
  Day 12 | -13.00 (4.813) | -14.38 (4.992)
  Day 13 | -12.15 (4.543) | -13.08 (6.873)
  Day 14 | -12.31 (4.309) | -14.38 (6.185)
  Day 15 | -12.08 (4.212) | -14.46 (5.592)
  Day 16 | -12.46 (3.597) | -15.00 (5.083)
  Day 17 | -12.31 (4.768) | -14.31 (5.721)
  Day 18 | -12.62 (4.753) | -14.15 (6.012)
  Day 19 | -12.62 (4.556) | -14.54 (5.577)
  Day 20: number analyzed (Participants) | 12 | 12
  Day 20 | -13.17 (3.810) | -15.83 (4.569)
  Day 21 | -11.77 (5.262) | -15.15 (5.535)
  Day 22 | -12.31 (4.404) | -15.08 (5.251)
  Day 23 | -11.92 (4.873) | -15.38 (5.091)
  Day 24 | -13.23 (4.419) | -15.69 (4.461)
  Day 25: number analyzed (Participants) | 12 | 13
  Day 25 | -14.83 (3.407) | -17.23 (4.850)
  Day 26 | -12.08 (4.645) | -15.08 (4.387)

11. Primary Outcome: Change From Baseline in Expired Air CO up to Day 26
Time Frame: Baseline, Days 4, 13, 17, 21, 26
Population: PD Set: All participants in the PK set who had an available baseline result and at least 1 on-treatment result with regards to urine cotinine, expired air CO or daily cigarette consumption and did not incur a major protocol deviation in a way that may have invalidated or biased the PD results.
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 13 | 13
ppm
  Day 4 | -13.2 (8.34) | -13.8 (7.03)
  Day 13: number analyzed (Participants) | 13 | 12
  Day 13 | -15.3 (8.02) | -15.9 (6.84)
  Day 17 | -16.0 (7.93) | -16.2 (5.81)
  Day 21 | -16.4 (7.79) | -16.5 (6.08)
  Day 26 | -17.2 (8.33) | -17.9 (6.75)

12. Primary Outcome: Number of Participants Who Ceased or Continued Smoking on Day 26
Description: A status of "ceased smoking" is defined as not having smoked any cigarettes for the past 24 hours on Day 26 and having an expired CO level <10 ppm on Day 26.
Time Frame: Day 26
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 13 | 13
Participants
  Ceased Smoking | 5 | 7
  Continued Smoking | 8 | 6

13. Primary Outcome: Change From Baseline Over Time in Urine Cotinine
Time Frame: Baseline, Days 4, 13, 17, 21, 26
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 13 | 13
ng/mL
  Day 4 | -1040.8 (579.78) | -1339.2 (550.74)
  Day 13 | -1010.0 (797.78) | -1309.3 (761.77)
  Day 17 | -1012.1 (710.39) | -1405.2 (814.08)
  Day 21 | -1095.1 (679.81) | -1446.3 (828.68)
  Day 26 | -1362.2 (545.84) | -1640.2 (688.84)

14. Primary Outcome: Change From Baseline Over Time in TCQ-SF Score: Emotionality
Description: The TCQ-SF is a 12-item questionnaire that assesses 4 components of tobacco craving: emotionality (3 items), expectancy (3 items), compulsivity (3 items) and purposefulness (3 items). Responses to each item are scored from 1 (strongly disagree) through 7 (strongly disagree). Component scores are defined as the sum of the scores within each component. The total score is defined as the sum of the 4 component scores. Emotionality scores may range from 3 to 21, with lower scores indicating weaker emotional signs of tobacco craving.
Time Frame: Baseline (Day -1), Days 4, 13, 17, 21, 26
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 13 | 13
score on a scale
  Day 4 | -5.2 (5.40) | -6.0 (5.03)
  Day 13 | -4.9 (5.96) | -7.2 (4.88)
  Day 17 | -5.8 (6.12) | -7.3 (5.06)
  Day 21 | -5.8 (6.38) | -7.6 (5.09)
  Day 26 | -5.7 (7.00) | -8.2 (4.98)

15. Primary Outcome: Change From Baseline Over Time in TCQ-SF Score: Expectancy
Description: The TCQ-SF is a 12-item questionnaire that assesses 4 components of tobacco craving: emotionality (3 items), expectancy (3 items), compulsivity (3 items) and purposefulness (3 items). Responses to each item are scored from 1 (strongly disagree) through 7 (strongly disagree). Component scores are defined as the sum of the scores within each component. The total score is defined as the sum of the 4 component scores. Expectancy scores may range from 3 to 21, with lower scores indicating less positive expectations about smoking.
Time Frame: Baseline (Day -1), Days 4, 13, 17, 21, 26
Population: PD Set: All participants in the PK set who had an available baseline result and at least 1 on-treatment result with regards to urine cotinine, expired air CO or daily cigarette consumption and did not incur a major protocol deviation in a way that may have invalidated or biased the PD results. Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 13 | 13
score on a scale
  Day 4: number analyzed (Participants) | 13 | 12
  Day 4 | -3.8 (5.89) | -8.0 (6.00)
  Day 13 | -3.5 (7.83) | -8.4 (5.91)
  Day 17 | -4.7 (6.96) | -8.8 (5.82)
  Day 21 | -5.2 (6.56) | -9.2 (5.75)
  Day 26 | -6.2 (6.40) | -9.8 (6.15)

16. Primary Outcome: Change From Baseline Over Time in TCQ-SF Score: Compulsivity
Description: The TCQ-SF is a 12-item questionnaire that assesses 4 components of tobacco craving: emotionality (3 items), expectancy (3 items), compulsivity (3 items) and purposefulness (3 items). Responses to each item are scored from 1 (strongly disagree) through 7 (strongly agree). Component scores are defined as the sum of the scores within each component. The total score is defined as the sum of the 4 component scores. Compulsivity scores may range from 3 to 21, with lower scores indicating compulsion to smoke was a lesser component of tobacco craving.
Time Frame: Baseline (Day -1), Days 4, 13, 17, 21, 26
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 13 | 13
score on a scale
  Day 4 | -3.2 (3.18) | -3.5 (4.74)
  Day 13 | -3.7 (6.56) | -4.9 (4.77)
  Day 17 | -4.4 (6.32) | -5.2 (4.44)
  Day 21 | -4.4 (5.49) | -5.3 (4.82)
  Day 26 | -4.3 (5.94) | -5.8 (4.59)

17. Primary Outcome: Change From Baseline Over Time in TCQ-SF Score: Purposefulness
Description: The TCQ-SF is a 12-item questionnaire that assesses 4 components of tobacco craving: emotionality (3 items), expectancy (3 items), compulsivity (3 items) and purposefulness (3 items). Responses to each item are scored from 1 (strongly disagree) through 7 (strongly disagree). Component scores are defined as the sum of the scores within each component. The total score is defined as the sum of the 4 component scores. Purposefulness scores may range from 3 to 21, with lower scores indicating stronger ability to not smoke.
Time Frame: Baseline (Day -1), Days 4, 13, 17, 21, 26
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 13 | 13
score on a scale
  Day 4 | -6.5 (2.93) | -7.5 (4.99)
  Day 13 | -6.6 (6.34) | -9.1 (5.45)
  Day 17 | -7.6 (6.33) | -9.2 (6.09)
  Day 21 | -7.8 (6.48) | -10.3 (5.65)
  Day 26 | -9.0 (5.15) | -11.1 (5.54)

18. Primary Outcome: Change From Baseline Over Time in TCQ-SF Score: Total Score
Description: The TCQ-SF is a 12-item questionnaire that assesses 4 components of tobacco craving: emotionality (3 items), expectancy (3 items), compulsivity (3 items) and purposefulness (3 items). Responses to each item are scored from 1 (strongly disagree) through 7 (strongly disagree). Component scores are defined as the sum of the scores within each component. The total score is defined as the sum of the 4 component scores. Total scores may range from 12 to 84, with lower scores indicating lower tobacco craving.
Time Frame: Baseline (Day -1), Days 4, 13, 17, 21, 26
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 13 | 13
score on a scale
  Day 4: number analyzed (Participants) | 13 | 12
  Day 4 | -18.7 (12.88) | -26.0 (16.06)
  Day 13 | -18.7 (22.11) | -29.6 (16.58)
  Day 17 | -22.5 (22.17) | -30.5 (16.51)
  Day 21 | -23.2 (21.79) | -32.5 (16.62)
  Day 26 | -25.2 (20.55) | -34.8 (16.85)

19. Secondary Outcome: Cytisine Amount Excreted in Urine Over Time (Ae0-24h)
Time Frame: Day 1 (6 times daily at 2-hour intervals); after the administration of the single dose of cytisine on Day 25
Population: PK Set: All randomized subjects who completed all cytisine dosing on Days 1-3, completed >90% cytisine dosing on Days 4-25 and complied with protocol-specified criteria.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 13 | 13
mg
  Day 1 | 7.95 (14.3) | 16.5 (12.0)
  Day 25 | 1.54 (17.4) | 3.14 (12.6)

20. Secondary Outcome: Percent of Drug Excreted in Urine (Ae%)
Time Frame: Day 1 (6 times daily at 2-hour intervals); after the administration of the single dose of cytisine on Day 25
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of excreted drug
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 13 | 13
percentage of excreted drug
  Day 1 | 88.3 (14.3) | 91.6 (12.0)
  Day 25 | 102 (17.4) | 105 (12.5)

21. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, and Discontinuation of Study Drug Due to TEAEs
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical trial subject administered a medicinal product and which does not necessarily have a causal relationship with the treatment. A serious adverse event (SAE) is defined as an AE that results in any of the following: results in death; is life-threatening; requires hospitalisation or prolongs existing inpatient's hospitalisation; results in persistent or significant disability or incapacity; results in a congenital abnormality or birth defect; is an important medical event which requires medical intervention to prevent any of the above outcomes.TEAEs are defined as AEs not present prior to first administration of investigational product, or AEs present before first administration of investigational product that worsen after the participant receives the first dose of investigational product.
Time Frame: From first dose of study drug through Day 26 plus 6-8 days
Population: Safety Set: all randomized participants who received at least one dose of cytisine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 13 | 13
Participants
  TEAEs | 9 | 9
  Serious TEAEs | 0 | 0
  Discontinuation of Study Drug due to TEAE | 0 | 0

22. Secondary Outcome: Number of Participants With Clinically Significant Values in Biochemistry, Hematology, and Urinalysis
Time Frame: up to Day 26
Population: Safety Set: all randomized participants who received at least one dose of cytisine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 13 | 13
Participants
  Biochemistry | 0 | 0
  Hematology | 0 | 0
  Urinalysis | 0 | 0

23. Secondary Outcome: Number of Participants With Clinically Significant Values in Vital Signs and Physical Examinations
Time Frame: up to Day 26
Population: Safety Set: all randomized participants who received at least one dose of cytisine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 13 | 13
Participants
  Vital Signs | 0 | 0
  Physical Examinations | 0 | 0

24. Secondary Outcome: Number of Participants With Clinically Significant Changes in 12-lead Electrocardiogram (ECG) Parameters
Time Frame: up to Day 26
Population: ECG Set: all participants who received at least 1 dose of cytisine, with at least 1 available baseline ECG and at least 1 on-treatment ECG.
Measure: Count of Participants; unit: Participants
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 13 | 13
Participants | 0 | 0

25. Secondary Outcome: Number of Participants With Holter ECG Outlier Values
Description: Based on the mean of the triplicate recordings at each time point. Increase (↑)/decrease (↓) calculated from Baseline (BL), defined as the mean of all recordings taken prior to dosing on Day 1 (i.e. -30 minutes and -15 minutes). A participant with multiple occurrences of an event is counted only once per event.
Time Frame: on Day 1 and Day 25 at 30 and 15 minutes prior to the first dose and 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours and 24 hours post dose
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
Number analyzed (Participants) | 13 | 13
Participants
  Day 1: Heart Rate <50 bpm & ↓ ≥ 25% | 0 | 0
  Day 1: Heart Rate >100 bpm & ↑ ≥25% | 1 | 0
  Day 1: PR Interval >200 mSec & ↑ ≥25% | 0 | 0
  Day 1: QRS Duration >100 mSec & ↑ ≥25% | 0 | 0
  Day 1: QT Interval >500 mSec & BL ≤500 mSec | 0 | 0
  Day 1: QTcF Interval >500 mSec & BL ≤500 mSec | 0 | 0
  Day 1: QTcF Interval >480 mSec & BL ≤480 mSec | 0 | 0
  Day 1: QTcF Interval >450 mSec & BL ≤450 mSec | 0 | 1
  Day 25: Heart Rate <50 bpm & ↓ ≥ 25% | 0 | 0
  Day 25: Heart Rate >100 bpm & ↑ ≥25% | 1 | 0
  Day 25: PR Interval >200 mSec & ↑ ≥25% | 0 | 0
  Day 25: QRS Duration >100 mSec & ↑ ≥25% | 0 | 1
  Day 25: QT Interval >500 mSec & BL ≤500 mSec | 0 | 0
  Day 25: QTcF Interval >500 mSec & BL ≤500 mSec | 0 | 0
  Day 25: QTcF Interval >480 mSec & BL ≤480 mSec | 0 | 0
  Day 25: QTcF Interval >450 mSec & BL ≤450 mSec | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug through Day 26 plus 6-8 days
Description: TEAEs are presented. TEAEs are defined as AEs not present prior to first administration of investigational product, or AEs present before first administration of investigational product that worsen after the participant receives the first dose of investigational product.
Arm/Group | Cytisine 1.5 mg | Cytisine 3.0 mg
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 9/13 | 9/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cytisine 1.5 mg (N=13) | Cytisine 3.0 mg (N=13)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Tooth loss (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 1
Chest discomfort (General disorders) | 0 | 1
Medical device site reaction (General disorders) | 1 | 1
Peripheral swelling (General disorders) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Headache (Nervous system disorders) | 4 | 6
Vision blurred (Nervous system disorders) | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinonasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are bound by requirements outlined in their individual clinical trial agreements with regard to publication of trial results.

DOCUMENTS (2):
  • Study Protocol (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/11/NCT03303911/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT03303911/SAP_001.pdf